CLINICAL TRIAL: NCT00002828
Title: PHASE I TRIAL OF SEQUENTIAL TOMUDEX AND 5-FLUOROURACIL IN SUBJECTS WITH ADVANCED COLORECTAL CARCINOMA
Brief Title: Chemotherapy With Raltitrexed and Fluorouracil in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 95-021; CDR0000065019 (Registry Identifier: PDQ (Physician Data Query)); ZENECA-MSKCC-95021A4; NCI-V96-0987
Record Dates: First submitted 1999-11-01; First posted 2003-11-24 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; raltitrexed

INTERVENTIONS:
Drug: fluorouracil
Drug: raltitrexed

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of raltitrexed and fluorouracil in treating patients who have colorectal cancer that is metastatic, recurrent, or cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of raltitrexed when administered with fluorouracil in patients with advanced colorectal carcinoma. II. Determine the toxicity and safety of this regimen in these patients. III. Assess, in a preliminary manner, the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of raltitrexed. Patients receive raltitrexed IV over 15 minutes followed 24 hours later by fluorouracil IV. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of raltitrexed until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose immediately preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6-10 patients are treated at the MTD. Patients are followed for 6 weeks.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 5-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic, locally recurrent, or surgically unresectable colorectal carcinoma Measurable disease No CNS metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2.5 times normal (5 times normal if known liver metastases) Renal: Creatinine no greater than 1.5 mg/dL Other: No severe concurrent infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 1 prior chemotherapy regimen Prior fluorouracil-based regimen for advanced colorectal cancer allowed Prior fluorouracil with radiotherapy not considered therapy for advanced disease At least 4 weeks since prior chemotherapy (8 weeks for mitomycin or nitrosoureas) and recovered Endocrine therapy: No concurrent steroids except for antiemesis or as replacement therapy Radiotherapy: See Chemotherapy No prior radiotherapy to more than 30% of bone marrow Surgery: See Disease Characteristics At least 4 weeks since prior surgery unless fully recovered Other: No concurrent vitamin supplements containing folic acid No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-04; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States